CLINICAL TRIAL: NCT05734716
Title: Colorado-Oregon Altitude Study
Acronym: COAST
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oregon (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY00000019
Record Dates: First submitted 2023-01-30; First posted 2023-02-21 (Actual); Last update posted 2023-03-10 (Actual); Status verified 2023-03

CONDITIONS: Acute Mountain Sickness
MeSH Terms: conditions — Altitude Sickness | interventions — Erythropoietin; Ferric Oxide, Saccharated

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Participants and researchers involved in data collection are blinded to the treatment assignment of all participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- EPO Arm (Experimental): participants administered subcutaneous erythropoietin injection (50 IU/kg 3x/week for 3 weeks) prior to ascent to altitutude. participants additionally administered sham intravenous treatment twice, with dosages occurring three weeks apart and final shame dose occurring 48 hours prior to ascent to altitude.
  Interventions: Drug: Erythropoietin
- Iron Arm (Experimental): participants administered intravenous iron sucrose (200mg) twice, dosages occurring three weeks apart with final dosing occurring 48 hours prior to ascent to altitude. Participants additionally administered sham subcutaneous injection (sterile saline) 3x/week for 3 weeks.
  Interventions: Drug: Iron sucrose (Venofer)
- Placebo (Placebo Comparator): participants administered sham injections (sterile saline) 3x/week for 3 weeks as well as sham intravenous infusion (sterile saline) twice with dosages occurring three weeks apart and final dosing occurring 48 hours prior to ascent to altitude.
  Interventions: Drug: Sterile Sodium Chloride

INTERVENTIONS:
Drug: Erythropoietin — use of erythropoietin to stimulate red blood cell development prior to ascent to altitude
  Arms: EPO Arm
Drug: Iron sucrose (Venofer) — use of iron sucrose to stimulate red blood cell development prior to ascent to altitude
  Arms: Iron Arm
Drug: Sterile Sodium Chloride — sham treatment with sterile saline
  Arms: Placebo

SUMMARY:
Investigating the utility of prophylactic treatment with iron sucrose and/or erythropoietin on the prevention of acute mountain sickness in fit, young, healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 40

Recreational athletes able to pass the APFTs

Men and women of any ethnic background

Medical and dental insurance

Able to read and speak English

Fully vaccinated against COVID-19

* If a subject is taking medication that is deemed safe and will not interfere with the main outcome measurements of the study as determined by clinical research staff, they will be included.
* If a subject had a previous mild to moderate COVID-19 infection but is deemed safe for all research activities by clinical research staff, then they will be included in the study.

Exclusion Criteria:

* Smokers

Previous severe COVID infection or contraction of any COVID infection occurring during the study. Previous mild to moderate COVID infections will be considered for the study on a case-by-case basis as determined safe by clinical research staff (see inclusion criteria).

Carboxyhemoglobin values (HbCO) 3% or greater at baseline

Diseases or disorders known to be affected by hypoxia or the drugs used in this study, including but not limited to hypotension, anemia, sickle cell trait or disease, and diabetes.

Anyone unable to receive the investigational drugs used in this protocol (EPO or iron).

Those with a history of significant head injury, migraines or seizures.

Anyone that is pregnant or trying to become pregnant.

Any medication determined by the clinical research staff to be unsafe or to interfere with the outcome measurements of the study.

Those with inability to be headache-free when consuming the amount of caffeine in two six-ounce cups of coffee or less per day.

Extended exposure (>6 hours) to high altitude above 1000m in the month leading up to departure to Colorado.

Those who have been on an airline flight over six hours (the lowered cabin pressure for an extended period of time approximates exposure to high altitude) within the month leading up to departure to Colorado.

Those who are unable to achieve the minimum physical criteria as outlined above.

Anyone with lung function below the lower limit of normal per GLI standards.

Previous diagnosis of high altitude pulmonary edema or high altitude cerebral edema upon altitude exposure.

Failure to get fully vaccinated against COVID-19. Choosing not to be vaccinated will result in exclusion.

Family history of clotting disorders, anemia or venous thrombosis.

Plans for professional competition during or within 1 week after participation in this study as participation may enhance your aerobic performance

Presence or absence of a PFO once we have enrolled a sufficient number of each group representation in the general population (e.g., ~40% of population has a PFO and ~60% does not). However, all subjects will be allowed to complete all baseline screening to assure that we will have enough subjects to go to Colorado

Biological sex once we have enrolled a sufficient number of males and/or females as we are aiming to enroll ~50% of each sex. However, all subjects will be allowed to complete all baseline screening to assure that we will have enough subjects to go to Colorado.

Subjects will be excluded from telemetric pill ONLY if they have a history of obstructive diseases of the gastrointestinal tract including diverticulosis, diverticulitis, inflammatory bowel disease, peptic ulcer disease, Crohn's disease, ulcerative colitis, or previous GI surgery.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Lake Louise Score | Pre-ascension to altitude
  Lake Louise Score of Acute Mountain Sickness symptoms
Lake Louise Score | Day 1 ascent to altitude
  Lake Louise Score of Acute Mountain Sickness symptoms
Lake Louise Score | 24 hours after ascent to altitude
  Lake Louise Score of Acute Mountain Sickness symptoms
Hemoglobin Mass | Pre-ascent to altitude
  total mass of hemoglobin in body
Hemoglobin Mass | Day 1 of Altitude
  total mass of hemoglobin in body
Hemoglobin Mass | Day 7 of Altitude
  total mass of hemoglobin in body
Hemoglobin Mass | Day 13 of Altitude
  total mass of hemoglobin in body
five kilometer run time trial | Pre-ascension to altitude
  time to cover 5 kilometers
five kilometer run time trial | Day 1 of Altitude
  time to cover 5 kilometers
five kilometer run time trial | Day 7 of Altitude
  time to cover 5 kilometers
five kilometer run time trial | Day 13 of Altitude
  time to cover 5 kilometers
p50 | Pre-ascension to altitude
  oxygen partial pressure point at which hemoglobin is 50% saturated with oxygen
p50 | Day 1 of Altitude
  oxygen partial pressure point at which hemoglobin is 50% saturated with oxygen
p50 | Day 7 of Altitude
  oxygen partial pressure point at which hemoglobin is 50% saturated with oxygen
p50 | Day 13 of Altitude
  oxygen partial pressure point at which hemoglobin is 50% saturated with oxygen
rucksack carry | Pre-ascent to altitude
  time to complete rucksack (35 pounds) course
rucksack carry | Day 2 of altitude
  time to complete rucksack (35 pounds) course
rucksack carry | Day 14 of altitude
  time to complete rucksack (35 pounds) course
pulmonary arterial systolic pressure | Pre-ascent to altitude
  highest pressure experienced in pulmonary vasculature during cardiac cycle
pulmonary arterial systolic pressure | day 1 ascent to altitude
  highest pressure experienced in pulmonary vasculature during cardiac cycle
pulmonary arterial systolic pressure | day 7 ascent to altitude
  highest pressure experienced in pulmonary vasculature during cardiac cycle
pulmonary arterial systolic pressure | day 13 ascent to altitude
  highest pressure experienced in pulmonary vasculature during cardiac cycle
hypercapnic ventilatory response | Pre-ascent to altitude
  level of end-tidal carbon dioxide which stimulates a ventilatory response
hypercapnic ventilatory response | Day 1 of Altitude
  level of end-tidal carbon dioxide which stimulates a ventilatory response
hypercapnic ventilatory response | Day 7 of Altitude
  level of end-tidal carbon dioxide which stimulates a ventilatory response
hypercapnic ventilatory response | Day 13 of Altitude
  level of end-tidal carbon dioxide which stimulates a ventilatory response
body core temperature | during 5k time trial pre-ascent to altitude
  body core temperature as measured by telemetric pill
body core temperature | during 5k time trial day 1 of Altitude
  body core temperature as measured by telemetric pill
body core temperature | during 5k time trial day 7 of Altitude
  body core temperature as measured by telemetric pill
body core temperature | during 5k time trial day 13 of Altitude
  body core temperature as measured by telemetric pill

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Colorado Mountain College, Leadville, Colorado
  - Cardiopulmonary and Respiratory Physiology Lab, Eugene, Oregon

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-02): https://cdn.clinicaltrials.gov/large-docs/16/NCT05734716/Prot_SAP_000.pdf
  • Informed Consent Form (2022-06-17): https://cdn.clinicaltrials.gov/large-docs/16/NCT05734716/ICF_001.pdf